CLINICAL TRIAL: NCT05385042
Title: Iron Supplementation and Immune Responses to Maternal Vaccination in Pregnant Women
Brief Title: Iron and Immune Response to Vaccine (IRONMUM)
Acronym: IRONMUM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HCR22001
Record Dates: First submitted 2022-03-24; First posted 2022-05-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Related
Keywords: Iron supplementation; Immune responses; Maternal vaccination
MeSH Terms: interventions — thiamine hydrochloride; Vitamin B 12

STUDY DESIGN:
Masking Description: This is a prospective open-label study in which both participants and investigators know the identity of the treatment and its dosage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-anaemic pregnant women (Other): 50 pregnant women who have normal haematocrit (not anaemic) at 12 weeks.
  Interventions: Dietary Supplement: Sangobion and Thiamine Hydrochloride
- Anaemic pregnant women (Other): 100 pregnant women who have haematocrit below 33% (equates to Hb 11g/dL) in first trimester (<14 weeks gestation) and below 30% (equates to Hb 10g/dL).
  Interventions: Dietary Supplement: Sangobion, Thiamine hydrochloride and Vitamin B12

INTERVENTIONS:
Dietary Supplement: Sangobion and Thiamine Hydrochloride — Prophylactic dietary supplements: 1 capsule of Sangobion + separate Thiamine Hydrochloride tablet 100mg per day for 12 weeks.
  Then non-anaemic pregnant women will continue with prophylactic nutritional supplements until delivery.
  Arms: Non-anaemic pregnant women
Dietary Supplement: Sangobion, Thiamine hydrochloride and Vitamin B12 — Treatment dietary supplements: 3 capsules of Sangobion + separate Thiamine Hydrochloride tablet 100mg, Vit B12 100mcg per day for 12 weeks.
  If experience a therapeutic increase of 3% Haematocrit within 28 days (responders), they will continue with prophylactic nutritional supplements until delivery.
  If no affect in Haematocrit level within 28 days (non-responders; defined by trimester of diagnosis), they will be investigated for their serum ferritin and if this is low (<15ng/mL) intravenous (iv) iron supplement (Venofer®) will be provided. The dose will be calculated for the individual concerned (required iron dose (mg) = (2.4 x (target Hb of 11g/dL (Ht 33%) x pre-pregnancy weight (kg) +1000mg for replenishment of stores). Doses will be administered by slow iv infusion 200 mg per dose (maximum of 3 doses per week).
  Following treatment they will continue with prophylactic nutritional supplements.
  Arms: Anaemic pregnant women

SUMMARY:
Iron deficiency causes anaemia and is common in pregnant women especially for those living in tropical regions where a high burden of infection and poor nutrition can compromise health. Low iron has been recognized as a cause of poor immune response because the group of cells that need to increase to make the immune response need iron to function. Vaccination is an important part of care during pregnancy because components of the immune response can cross the placenta and protect the young infant. More recently COVID-19 vaccination has also been recommended for pregnant women due to their higher risk of dying from this infection. Deeper investigation of whether low iron results in poor immune response is needed because the vaccines may not be providing as much protection as needed. The World Health Organization also recommends nutritional iron supplements in pregnancy and whether these improve immune response to vaccines is also not known. This study aims to test the body's immune response to recommended vaccines in pregnant women (tetanus and diphtheria (combination) and COVID-19 vaccine (if indicated)) who are anaemic and receiving iron supplements and compare their response to women who are not anaemic, who only receive a preventive, lower dose of supplement.

DETAILED DESCRIPTION:
This is a prospective interventional open label cohort study with an exploratory framework. After assessment of gestation by routine ultrasound, women will be invited to participate if they have a viable, singleton pregnancy with a gestation < 28 weeks. Consenting pregnant women will be enrolled at first antenatal clinic [7] visit and receive tetanus and diphtheria immunisation after confirmation of vaccination history, and SARS-CoV-2 immunisation (first dose if indicated). All women will be classified as non-anaemic or anaemic based on haematocrit (Haematocrit<33% in first trimester (defined <14 weeks) and Haematocrit <30% in 2nd trimester (defined 14 to <28 weeks)). Women will be assigned to groups and receive prophylactic (non-anaemic) or treatment (anaemic) doses of nutritional supplements, respectively, as per routine practice. These supplements will be provided daily for 3 months (12 weeks) and women will be followed up at day 7, 1 month (day 28), 2 and 3 months. There after they will follow routine antenatal care until birth when a cord blood sample will be taken. Mother and infant blood samples will be taken at the 2 months post-partum visit when the newborn attends for routine vaccinations of the expanded program of immunisation. Immunological and haematological responses will be measured by venous blood sampling and finger-prick sampling (routine at the clinics) at study visits; as will adverse events in relation to nutritional supplements by monthly questions using a checklist of common reactions to oral iron. The Adherence Starts with Knowledge (ASK-12) instrument has been modified and used in this population and will be compared to the Haematocrit levels, the pill count and adverse events, as a measure of adherence.

IRONMUM study is funded by Procter and Gamble. The grant reference number is Thailand-UK-IRONMUM-2021-01.

ELIGIBILITY:
Inclusion Criteria:

1. Viable singleton pregnancy<28 weeks confirmed by ultrasound
2. 18 years and older
3. Willingness and ability to comply with the study protocol for the duration of the study
4. Can understand information about the study and provide consent

Exclusion Criteria:

1. Any diphtheria-tetanus vaccine within the previous 2 years
2. History of allergic reaction to diphtheria-tetanus or COVID-19 vaccine
3. Haematocrit <21% or Haematocrit >50%
4. Known severe haemoglobinopathy (HbE/beta-thalassaemia syndrome, beta-thalassaemia major or HbH syndrome)* or G6PD deficiency

   * Iron supplementation is safe in pregnant women with haemoglobin E, alpha-thalassemia 1, or beta-thalassemia carriers.
5. HIV-positive
6. Slide confirmed presence of malaria
7. Fever (defined at >37.5°C)
8. Symptoms of COVID (these women will be PCR tested as routine in clinic)
9. Known severe medical or obstetric complication e.g. valvular heart disease, placenta praevia
10. Known or clinical vitB12 deficiency as indicated by megaloblastic anaemia (pernicious anaemia or clinical symptoms)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 150 (Estimated)
Dates: Start 2022-06-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Antibody responses to maternal vaccine | change from baseline before immunisation and at 7-days and 28-days after immunisation, and at 2 months post-partum in mother and infant.
  Antibody responses to diphtheria-tetanus and SARS-CoV-2 immunisation, measured by ELISA.

SECONDARY OUTCOMES:
Cellular Immune response post-immunisation measured by Mass Cytometry (plasma cells and circulating T-follicular helper cells). | 7-days after immunisation
Profile of the circulating immune system components over the course of pregnancy measured by CyTOF | change from before immunisation, 7-days and 28-days after immunization and until 2 months post-partum in mother and infant
Haematological, iron and inflammatory parameters including: Hb, MCV, haematocrit serum iron, ferritin, TSAT, hepcidin, CRP, G6PD, Hb typing. | change from before immunisation, 7-days and 28-days after immunization and at 2 months post-partum in mother and infant
Haematocrit from baseline if anaemic at baseline according to trimester of gestation | change from baseline and month 1,2 and 3, and delivery
Modified Adherence Starts with Knowledge (ASK-12) questionnaire including pill count. | Month 1,2 and 3
  ASK-12 scores can range from 12-60, with higher scores representing greater barriers to adherence]
To monitor safety of iron supplements | change from baseline and month 1,2 and 3
  Monitor adverse events in mother and neonate - gastrointestinal (e.g. constipation, diarrhea, infection)

OTHER OUTCOMES:
To assess if the amount of betel nut consumption relates to Haematocrit response | change from baseline and month 1,2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Hal Drakesmith, Dr., Principal Investigator — MRC Human Immunology Unit, John Radcliffe Hospital, University of Oxford, OX3 9DS UK
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All personal details of participants will be de-identified. These data including laboratory investigation results will be stored and may be shared to other researchers to apply in their research in accordance with the MORU data sharing policy.
Time Frame: After completion of trial activities. PI will upload results within 12 months of the end of the trial declaration.
Access Criteria: MORU Data Sharing Policy. The criteria for authorship will be consistent with the international guidelines (http://www.icmje.org/#author).
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing